CLINICAL TRIAL: NCT03838250
Title: A Phase I, Open-Label, Single-Dose Study to Evaluate the Safety and Efficacy of Hepatic Artery Injection of Autologous Human Bone Marrow-Derived Mesenchymal Stem Cells (Cellgram™) in Patients With Alcoholic Liver Cirrhosis
Brief Title: Study to Evaluate Hepatic Artery Injection of Autologous Human Bone Marrow-Derived MSCs in Patients With Alcoholic LC
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pharmicell Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PMC-P-08
Record Dates: First submitted 2019-01-07; First posted 2019-02-12 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Alcoholic Liver Cirrhosis
Keywords: Alcoholic; Liver; Cirrhosis; Liver Disease
MeSH Terms: conditions — Liver Cirrhosis, Alcoholic; Fibrosis; Liver Diseases

STUDY DESIGN:
Intervention Model Description: A single-dose injection of autologous bone marrow-derived mesenchymal stem cells (Cellgram™) will be administered to the patient by an experienced interventional radiologist.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cellgram™ (Bone marrow-derived MSCs) (Experimental): Infusion Cellgram™(Bone marrow-derived MSCs). Single dose administration of approximately 5 x 10^7 cells/10 mL (range: 4.5 x 10^7 to 5.5 x 10^7 cells/10 mL) via the hepatic artery.
  Interventions: Biological: Cellgram™ (Bone marrow-derived MSCs)

INTERVENTIONS:
Biological: Cellgram™ (Bone marrow-derived MSCs) — Approximately 15 to 30 mL of bone marrow is aspirated from the posterior iliac crest of patients under local anesthesia. Approximately 30 days (±7 days) after BM aspiration, the participant will return to the study center for admission and for the infusion Cellgram™ (Bone marrow-derived MSCs).

SUMMARY:
This study is to evaluate the safety and efficacy of a single dose of Cellgram™ delivered via hepatic artery in patients with decompensated alcoholic liver cirrhosis.

DETAILED DESCRIPTION:
After providing written informed consent, subjects will return to the study center for further evaluation and to have their Bone marrow harvested by an experienced hematologist or interventional radiologist.

Within approximately 1 month (30 ± 7 days) after Bone marrow aspiration, study participants will be admitted to the study center on Day 1.

At the study center, the participant will undergo hepatic artery catheterization by an interventional radiologist who will inject a single dose of Cellgram™. Participants will remain as in-patients and be observed for 24 hours post-infusion. Following discharge, participants will periodically return to the study center for study assessment visits over a period of 1 year.

When a suitable candidate is identified by the Investigator, the Investigator or designated healthcare professional will ask the patient about his/her willingness to be included in the clinical study. Following this, patients will be allowed sufficient time, in their own opinion, to consider study entry, and will be offered the opportunity to ask any further questions prior to signing the informed consent form.

ELIGIBILITY:
Inclusion Criteria:

1. Alcoholic liver cirrhosis as diagnosed by clinical, biochemical, radiological, or histological evidence.
2. Male or female, 18 to 70 years of age, inclusive.
3. Child-Pugh class B (7 to 9 points)
4. Capable, in the Investigators opinion, of undergoing hepatic artery catheterization.
5. No consumption of alcohol or other potentially hepatotoxic substances considered clinically relevant in the opinion of the Investigator, within 6 months prior to screening and throughout the study.
6. Provision of informed consent by the patient (or their legal representative) to participate in the clinical study.
7. Able, in the Investigator's opinion, to comply with the requirements of the protocol (including the follow-up period).
8. Females of childbearing potential must test negative on standard urine pregnancy test and must be willing to practice appropriate contraceptive methods for the duration of the study. Highly effective methods of birth control include hormonal birth control, intrauterine devices (IUDs), or any double-barrier method (sponges, female condoms) used by the woman in addition to contraception used by their male partner such as vasectomy or condom supplemented with spermicide.

Exclusion Criteria:

1. Current diagnosis of malignant hematologic disease (e.g., acute myeloid leukemia, acute lymphoblastic leukemia, non-Hodgkin's lymphoma, Hodgkin's lymphoma, multiple myeloma).
2. Etiology other than alcohol for underlying liver cirrhosis.
3. Baseline creatinine >1.7 mg/dL and/or estimated glomerular filtration rate (eGFR) <30 mL/min/1.73 m2
4. Clinical history of a solid cancer within 5 years prior to screening or current diagnosis of a solid cancer (including hepatocellular carcinoma assessed by ultrasonography and elevated AFP level) and currently receiving cancer treatment.

   Continuous use of a clinically relevant amount of steroids or antibiotics within 1 month prior to screening. Clinical relevance will be determined by the Investigator.
5. Model for End-Stage Liver Disease score >20.
6. International normalized ratio >3.0 and/or platelet counts <30,000/mm3
7. Major operation within 3 months prior to screening.
8. Presence of extrahepatic biliary stricture.
9. Participant has undergone transjugular intrahepatic portosystemic shunt.
10. Active hepatic artery or portal vein thrombosis.
11. Presence of advanced hepatic encephalopathy Stages 3-4 (West Haven criteria) at the time of screening.
12. Active variceal bleeding during the last 6 months before screening.
13. Severe cardiac, renal, or respiratory failure.
14. Positive serological test results for human immunodeficiency virus (HIV), HCV, hepatitis B surface antigen (HBsAg) and/or syphilis.
15. Patient is pregnant or breast feeding, or planning to become pregnant while enrolled in the study, up to the EOS visit.
16. Positive urine pregnancy test at Screening.
17. Drug abuse within the past 2 years (as confirmed by patient disclosure or a urine drug screen conducted at Screening).
18. Participation in an interventional clinical study within 30 days prior to screening.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-06-20 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of Serious Adverse Events | 12 months
  An SAE suggests a significant hazard, contraindication, side-effect, or precaution. With respect to human clinical experience, this includes any event that:
  * Results in death.
  * Is life-threatening.*
  * Requires in-patient hospitalization or prolongation of existing hospitalization.
  * Results in persistent or significant disability/incapacity.
  * Is a congenital anomaly/birth defect.
  * Other medically important condition
    * Life-threatening in the definition of a SAE or adverse reaction refers to an event in which the patient was at risk of death at the time of event; it does not refer to an event, which hypothetically might have caused death if it were more severe.

SECONDARY OUTCOMES:
Number of patients with Hepatocellular carcinoma (primary liver cancer) development | 12 months
  assessed via ultrasonography and alpha fetoprotein [AFP] analysis
Incidence of Adverse Events | 12 months
  Incidence of Adverse Events as assessed by vital signs, physical examination, safety laboratory tests, and patient reporting
Liver stiffness measurement | 12 months
  with transient elastography (i.e., FibroScan®)
How well the Liver is functioning | 12 months
  by tests including: serum levels of aspartate aminotransferase (AST), alanine aminotransferase (ALT), bilirubin, albumin, gamma glutamyl transpeptidase (GGT) and creatinine.
  Units of Measure: AST will be report in U/L. ALT will be report in U/L. GGT will be report in U/L. Bilirubin will be report in mg/dL. creatinine will be report in mg/dL. Albumin will be report in g/dL
Chronic liver disease as assessed by the Child-Pugh score | 12 months
  The Child-Pugh Score will be used to determine the prognosis, required strength of treatment and the necessity of liver transplantation. The score employs 5 clinical measures of liver disease (total bilirubin, serum albumin, INR, ascites and hepatic encephalopathy). Each parameter is scored 1 to 3, with 3 indicating the most severe derangement.
Model for End-Stage Liver Disease (MELD) Score | 12 months
  MELD uses the patient's values for serum bilirubin, serum creatinine, and the INR for PT to predict survival. It is calculated according to the following formula defined by Kamath et al (2001):
  MELD = 3.78×ln[serum bilirubin (mg/dL)] + 11.2×ln[INR] + 9.57×ln[serum creatinine (mg/dL)] + 6.43
Overall survival | 12 months
  defined as the time from infusion until death from any cause during the study period.
Quality of life as assessed by 36-Item Short Form Survey (SF-36) Questionnaire | 12 months
  The Short Form-36 Quality Of Life questionnaire will be recorded for each patient. The 8 subscales of the SF-36 (Physical Functioning, Role Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role Emotional, Mental Health) and 2 summary component measures (Physical Component Summary, Mental Component Summary) will be calculated and summarized.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Gallegos-Orozco, Ph.D, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Undecided